CLINICAL TRIAL: NCT04879355
Title: The Use of Spinal Needles for Ultrasound-guided Fine Needle Aspiration From Thyroid Nodules - a Protocol for a Multicentre Randomised Controlled Trial
Brief Title: Spinal Needles in Ultrasound-guided Fine Needle Aspirations From Thyroid Nodules
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Preben Homøe (Other)
Collaborators: Herlev Hospital (Other); Rigshospitalet, Denmark (Other)
Responsible Party: Sponsor-Investigator, Preben Homøe, Professor, Zealand University Hospital
Organization: Zealand University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: SJ-878
Record Dates: First submitted 2021-03-07; First posted 2021-05-10 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2022-06

CONDITIONS: Thyroid Nodule
MeSH Terms: conditions — Thyroid Nodule

STUDY DESIGN:
Intervention Model Description: Eligible patients are randomised at a 1:1-ratio to one of two parallel groups, and all patients are included in the analysis on an intention-to-treat basis.
Who Masked: Participant, Outcomes Assessor
Masking Description: The patients and the pathologists are blinded to the intervention, while the clinicians performing the FNAs are not.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Spinal needle (Experimental): Fine needle aspiration from thyroid nodules using af spinal needle.
  Interventions: Device: Spinal needle (25G)
- Conventional fine needle (Active Comparator): Fine needle aspiration from thyroid nodules using af conventional fine needle, which is traditionally used.
  Interventions: Device: Conventional fine needle (25G)

INTERVENTIONS:
Device: Spinal needle (25G) — Fine needle aspiration from thyroid nodules using a 25G spinal needle.
  Arms: Spinal needle
Device: Conventional fine needle (25G) — Fine needle aspiration from thyroid nodules using a conventional 25G fine needle
  Arms: Conventional fine needle

SUMMARY:
This is a multicentre, two-arm, randomised and controlled trial. Adults with thyroid nodules suspected of malignancy are to be included consecutively. A total of 350 patients are randomly assigned 1:1 to have FNA with a spinal (25G) or a conventional (25G) needle. The primary outcome is the rate of diagnostic cytological samples according to the Bethesda system. Secondary outcomes are diagnostic accuracy, patient's experienced pain and complication rates.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years of age.
2. Patients referred for evaluation of a cold nodule on thyroid scintigraphy and with EU-TIRADS score of 3 or higher.

   * Score 3 and > 20 mm in size.
   * Score 4 and >15 mm in size.
   * Score 5 and >10 mm in size.
3. Clinical suspicion of thyroid cancer:

   * PET-positive thyroid tumor.
   * Thyroid tumor and palsy of the recurrent laryngeal nerve.
   * Rapidly growing thyroid tumor.
   * Hard and/or immobile thyroid tumor.
   * Tumor in the thyroid with suspicious lymph nodes.

Exclusion Criteria:

* Previous participation in the study.
* Language or other barriers not allowing adequate information.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic rate | 1 year
  The percentage of samples evaluated as "diagnostic" by the pathologist.

SECONDARY OUTCOMES:
Complication rate | Till 1 month after last inclusion. Corresponding to about 1 year
  Complications, such as infections, bleedings or hematomas requiring treatment or admission, recurrent nerve injury and Horner's syndrome, will be recorded during the procedure. All patients are instructed to contact the department responsible for their management if they suspect complications. These will then be documented in the patient's medical record. At the end of the study period, the patient's medical records will be reviewed for admissions or contacts concerning complications.
Pain assessment | About 2 years
  Pain is assessed using the VAS (Visual Analog Scale) immediate after the procedure.
  The score is ranging from 0 to 10 with higher numbers indicating a more painful procedure.
Diagnostic accuracy | About 2 years
  Cytology from FNAB is compared with histology in the subgroup of patients who undergo surgery during the course of the study

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Andersen, MD, Principal Investigator — Zealand University Hospital, Køge, Denmark.
Locations (1):
- Zealand University Hospital, Koege, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Data collected in this trial can be shared upon request from other researchers after publication.
Supporting Information: Study Protocol, ICF, CSR

REFERENCES:
- [Derived] Andersen TV, Bennedbaek FN, Pedersen J, Rosenorn MR, Kiss K, Lelkaitis G, Andersen L, Hegedus L, Lomholt AF, Hahn CH, Hvilsom GB, Homoe P, Todsen T. Spinal versus conventional fine needle for ultrasound-guided thyroid nodule biopsy: a protocol for a randomised clinical trial. Dan Med J. 2022 Jul 21;69(8):A03220165. PMID 35959834